CLINICAL TRIAL: NCT04682860
Title: Management of Abdominal Pain in Acute Gastroenteritis Patients With Hyoscine Butylbromide: Randomized Double Blind Placebo Controlled Trial
Brief Title: Management of Abdominal Pain in Acute Gastroenteritis Patients With Hyoscine Butylbromide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Cagdas Yildirim, Ass. Prof., Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Çağdaş Yıldırım
Record Dates: First submitted 2020-12-14; First posted 2020-12-24 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Acute Gastroenteritis; Abdominal Pain
MeSH Terms: conditions — Abdominal Pain | interventions — Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): In the placebo arm, patients will be slowly injected with 2 ml of normal saline within 30 seconds
  Interventions: Other: Placebo
- Hyoscine N butylbromide (Active Comparator): In the treatment arm, the patient will be injected intravenously with 1ml 20 mg of Hyoscine butylbromide and 1 ml of normal saline intravenously within 30 seconds.
  Interventions: Drug: Hyoscine N Butylbromide

INTERVENTIONS:
Drug: Hyoscine N Butylbromide — Hyoscine N butylbromide injection for the treatment of abdominal pain in acute gastroenteritis
  Arms: Hyoscine N butylbromide
Other: Placebo — 2 ml of normal saline injection as placebo
  Arms: Placebo

SUMMARY:
One of the most common complaints of admission to the emergency room is gastroenteritis. One of the most common complaints in acute gastroenteritis is abdominal pain. The aim of our study is to investigate whether hyoscine butylbromide used within the indication has an effect on abdominal pain due to acute gastroenteritis. The main purpose of our study is to reduce the pain of the patient at 30th and 60th minutes compared to 0th minute.

ELIGIBILITY:
Inclusion Criteria:

* Patients with watery stools starting in the last 2 weeks and 3 times in 24 hours and abdominal pain

Exclusion Criteria:

* Peritonitis
* Hemodynamic instability
* Pregnancy
* Inability to give consent
* Medication given in the emergency room before being included in the study
* Taking pain medication within 4 hours
* Diabetes Mellitus and other neuropathic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
Pain Change | 30 minute and1 hour
  Pain change after intervention at 30th and 60th minute. Pain will assesed with Visual Analog Scale (100 mm). 13 mm of change at Visual Analog Scale will assesed as clinically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Çağdaş Yıldırım, Ass. Prof, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD maybe shared upon request

REFERENCES:
- [Background] Remington-Hobbs J, Petts G, Harris T. Emergency department management of undifferentiated abdominal pain with hyoscine butylbromide and paracetamol: a randomised control trial. Emerg Med J. 2012 Dec;29(12):989-94. doi: 10.1136/emermed-2011-200474. Epub 2012 Feb 3. PMID 22307926
- [Background] Arena C, Amoros JP, Vaillant V, Ambert-Balay K, Chikhi-Brachet R, Jourdan-Da Silva N, Varesi L, Arrighi J, Souty C, Blanchon T, Falchi A, Hanslik T. Acute diarrhea in adults consulting a general practitioner in France during winter: incidence, clinical characteristics, management and risk factors. BMC Infect Dis. 2014 Oct 30;14:574. doi: 10.1186/s12879-014-0574-4. PMID 25358721
- [Background] Shane AL, Mody RK, Crump JA, Tarr PI, Steiner TS, Kotloff K, Langley JM, Wanke C, Warren CA, Cheng AC, Cantey J, Pickering LK. 2017 Infectious Diseases Society of America Clinical Practice Guidelines for the Diagnosis and Management of Infectious Diarrhea. Clin Infect Dis. 2017 Nov 29;65(12):1963-1973. doi: 10.1093/cid/cix959. PMID 29194529